CLINICAL TRIAL: NCT02306304
Title: Ultra-sound for AAA Screening in Smoking Israeli Arab Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clalit Health Services (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Dr. Asaf Rabin, M.D., Clalit Health Services
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ClalitHS
Record Dates: First submitted 2014-11-26; First posted 2014-12-03 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Abdominal Aortic Aneurysm (AAA)
Keywords: Abdominal aortic aneurysm; Abdominal aortic aneurism; AAA; Screening; duplex ultra sound; Israeli Arab men; family physician
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Israeli Arab men (Other): Single arm study. The arm includes all enrolled patients screened by duplex ultra sound for abdominal aortic aneurysms.
  Interventions: Other: Duplex ultra sound screening for abdominal aortic aneurysms

INTERVENTIONS:
Other: Duplex ultra sound screening for abdominal aortic aneurysms — Duplex ultra sound screening for abdominal aortic aneurysms in Israeli Arab men, smokers or past smokers at the age of 60-80 years.

SUMMARY:
The study aims at screening Israeli Arab men, smokers or past smokers, for abdominal aortic aneurysms (AAA).

The screening is to be performed at the family doctors clinics in the rural arab erea of the north of Israel.

Goals:

The investigators aim at revealing the actual prevalence of AAA in the Israeli Arab smoking men population. By revealing this prevalence we believe the need for a nation-wide screening program for AAA will turn available for assessment.

In addition, the goal of improving the accessibility of health services for the Israeli Arab population is a key issue in the design of the research.

2000 patients are to be enrolled in the study over a period of 2 years. Each of the patients will be examined once for a duplex ultra-sound and will be classified into one of 4 sub-groups according to the maximal aortic diameter found.

DETAILED DESCRIPTION:
Study Protocol No.:0017-14-COM

Ultra-sound for AAA screening in smoking Israeli Arab men

Initiator & Head researcher:

Asaf Rabin, M.D. Vascular Clinic, Haifa and Western Galilee district, Clalit Health Services Horev Center, Haifa asafrabin@gmail.com

+972-527-950-905

Signature:

Contents

1. Study Rationale & References --------------------------- 4-5
2. Goals ----------------------------------------------------------- 6
3. Research Design ---------------------------------------------- 7
4. Inclusion and exclusion criteria ----------------------------- 8
5. CRF---------------------------------------------------------- 9-10
6. End Points & Follow up chart -------------------------- 11-12
7. Confidentiality ------------------------------------------------ 13

Study Rationale

In the United States ruptured abdominal aortic aneurysms (AAA) are the 15th leading cause of death overall and the 10th leading cause of death in men older than 55 years. The prevalence of AAA found in population-based ultrasonography (US) screening studies from various countries is about 4-9% in men and 1% in women older than 65yr.

If left untreated, the aneurysm continues to expand; thinning of the aortic wall ensues and rupture may eventually occur. Most of large AAA are asymptomatic and often rupture occurs with no warning signs.

Mortality due to rupture of an aortic aneurysm is high (80-90%), compared to 5-7% in elective surgery for AAA repair and even lower when treated by endovascular means (1-2%).

Ultra-sound can reliably demonstrate the aorta in 99% of the population, and its sensitivity and specificity in diagnosing AAA approaches 95-100%. Screening with Ultra-sound for AAA has been proved in multiple studies to reduce AAA related mortality by an average of 42% in the screened population compared with the non-screened population. The reduction in mortality was achieved in a cost effective way. Based on such studies a number of screening programs have been implemented in the United Kingdom (UK), United States (USA), Scotland and Sweden.

As for today there is no screening program for AAA in Israel. The investigators would like to conduct a study in a specific group of the population demonstrating the need for screening in such group.

The major risk factors for AAA include Age (>65 years), male gender and a history of ever smoking. It has been demonstrated that smoking rates among Israeli Arab men are significantly higher than those of Israeli Jewish men. Most of the Israeli Arab population inhabits rural areas with less access to hospitals and medical centers.

Therefore, the investigators decided to conduct a prospective study in which Israeli Arab men between the ages 60-80 years old, with a history of smoking, will undergo an ultra-sound examination for screening for AAA.

Goals The investigators aim at revealing the actual prevalence of AAA in the Israeli Arab smoking men population. By revealing this prevalence the investigators believe the need for a nation-wide screening program for AAA will turn available for assessment.

In addition, the goal of improving the accessibility of health services for the Israeli Arab population is a key issue in the design of the research. Performing the screening ultra-sound in the family-physician's clinics (see below under "Research Design") will save the patients the time and the trouble involved with being examined in the central vascular clinics. It will also improve the knowledge and awareness of the population in general and of the family-physicians in particular of the AAA disease and for the need of early diagnosis and treatment as mentioned above.

Last but not least, the private benefit of each patient either from ruling out the option of having an AAA or from diagnosis of an AAA and referral to treatment is a valuable by-product of the research.

Research Design 2000 men (according to the inclusion criteria) are planned to be included in the "screening study" over a period of one year to two years.

The family-physicians of the Haifa and Western Galilee district, Clalit Health Services will be notified by the head researcher about the research. The organization will be asked to provide a list of potential patients according to the inclusion and exclusion criteria. The list will only include patients whom the physician had addressed and whom had given their approval for being approached by the research team.

The patients will then be invited for a meeting with one of the researchers at the family-physician clinic. After a full explanation will be given, an informed consent form will be signed by the patient. Each patient will be documented on a Case Report Form (CRF) and will be given a code for the rest of the research. The coding system is aimed at securing the confidentiality of the patients' personal and medical information.

Then after, with the help of the technician a Duplex Ultra-sound examination of the abdominal aorta will be performed. Since the examination is performed after a 6 hours fasting period, the fasting instruction will be given to the patients in advance. The results of the scans will be recorded in each patient Case Report Form (CRF).

The patient will be classified according to the Duplex US findings into one of 4 sub-groups as detailed under "End-Points". A recommendation for further follow-up or treatment will be given to each patient and will be documented in his CRF accordingly. The results of the scan and the recommendations will be sent the patient and to his family-physician within a short period following the exam.

It is to be made clear both hereby and in the informed consent form that the consent of the patient to participate in the research bares no further obligations to follow the recommendations of the research team nor to be followed-up or treated under the umbrella of the vascular service of Haifa and Western Galilee district, Clalit Health Services.

Non-the-less, each of the patients is entitled for full follow-up and treatment by the vascular service of Haifa and Western Galilee district, Clalit Health Services regardless of his consent to participate in the research or to follow the research team recommendations.

Each patient will be documented digitally in a separate research file. A copy of the informed consent will be given to patient. The same document will be scanned and filed in the patients research file. The file will also contain the CRF and the exam results.

Study name: US for AAA screening in smoking Israeli Arab men

Patient code:

Date:

Place:

Case Report Form (CRF) Form filled at enrollment

1. Age (60-80):
2. Smoking:

   1. Active / in Past / No
   2. Y.P. -
3. Israeli Arab man: Yes / No
4. A known AAA
5. Previous operations of the abdominal aorta
6. Previous imaging study within the last 12 months, ruling-out AAA.
7. Match to inclusion criteria: Yes / No

   ---------------------------------------------------------------------------------
8. Weight:
9. Height:
10. Hypertension: Yes / No
11. Diabetes mellitus: Yes / No
12. Hypercholesterolemia/hyperlipidemia: Yes/ No
13. Ischemic heart disease:

    1. Myocardial infarction- Yes/ No
    2. Coronary artery bypass- Yes/ No
    3. Catheterization - Yes/ No
14. Origin of medical information:

    1. The patient - Yes / No
    2. The patient's relatives - Yes / No
    3. The patient's general physician - Yes / No
    4. Computerized medical file - Yes / No
    5. Other medical documents - Yes / No
15. Ultra-sound results:

    1. Abdominal aorta maximal diameter- _____ cm
    2. Sub-group - A / B / C / D

Date: ________ Physician name & signature:__________

End-Points & Follow up chart A formal report will be produced for every examination and will be signed by a vascular surgeon and sent to the patient and to his family-physician.

The examined patient will be classified into one of the listed sub-groups according to the measured maximal aortic diameter.

The head researcher will be responsible for inviting the patient for further follow-up or for additional work-up and treatment according to the findings.

Result of screening US:

* Sub-group A:

  * Normal Aorta (<3 cm)
  * No need for follow up or extra imaging
* Sub-group B:

  * Aortic Diameter ( 3-4.5 cm)
  * Needs follow up: Annual aortic US
* Sub-group C:

  * Aortic Diameter ( 4.5-5.5 cm)
  * Needs follow up: Semiannual aortic US
* Sub-group D:

  * Aortic Diameter (> 5.5cm)
  * Further investigation and treatment: referral to Vascular Surgeon for treatment.

Confidentiality

The head researcher is committed for the confidentiality of the personal and medical information of the patient participating in the research.

All the research documents will be coded and will contain no personal data. If personal details will be needed for the research they would be coded through a scrambling system for prevention of any identifying potential.

The research data will be saved on a stand-alone computer and raw data will not be transferred or shared via internet.

Clalit Health Services will be notified by the head-researcher for any occasion of data loss, theft or damage.

The head-researcher will share the research raw data with any 3rd party only after a clear approval of Clalit Health Services is obtained.

The research raw data will only be saved on a desk-top computer and not on any mobile electronic device.

ELIGIBILITY:
Inclusion Criteria:

* Arab men
* Age : 60-80 years old
* History of smoking

Exclusion Criteria:

* A known AAA
* Previous operations of the abdominal aorta
* Previous imaging study within the last 12 months, ruling-out AAA.

Ages: 60 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 913 (Actual)
Dates: Start 2015-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Abdominal aortic aneurysm prevalence in the represented population | 2 years
  At the end of enrollment, estimated time - 2 years, the prevalence will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Asaf Rabin, M.D., Principal Investigator — Clalit Heath Services
Locations (1):
- Clalit Health Services primary clinics, Haifa, Haifa and Western Galilee District & Northen District, Israel

REFERENCES:
- [Background] Fleming C, Whitlock EP, Beil TL, Lederle FA. Screening for abdominal aortic aneurysm: a best-evidence systematic review for the U.S. Preventive Services Task Force. Ann Intern Med. 2005 Feb 1;142(3):203-11. doi: 10.7326/0003-4819-142-3-200502010-00012. PMID 15684209
- [Background] Thompson SG, Ashton HA, Gao L, Buxton MJ, Scott RA; Multicentre Aneurysm Screening Study (MASS) Group. Final follow-up of the Multicentre Aneurysm Screening Study (MASS) randomized trial of abdominal aortic aneurysm screening. Br J Surg. 2012 Dec;99(12):1649-56. doi: 10.1002/bjs.8897. Epub 2012 Oct 3. PMID 23034729
- [Background] U.S. Preventive Services Task Force. Screening for abdominal aortic aneurysm: recommendation statement. Ann Intern Med. 2005 Feb 1;142(3):198-202. doi: 10.7326/0003-4819-142-3-200502010-00011. No abstract available. PMID 15684208
- [Background] Norman PE, Jamrozik K, Lawrence-Brown MM, Le MT, Spencer CA, Tuohy RJ, Parsons RW, Dickinson JA. Population based randomised controlled trial on impact of screening on mortality from abdominal aortic aneurysm. BMJ. 2004 Nov 27;329(7477):1259. doi: 10.1136/bmj.38272.478438.55. Epub 2004 Nov 15. PMID 15545293
- [Background] Wilmink AB, Quick CR, Hubbard CS, Day NE. Effectiveness and cost of screening for abdominal aortic aneurysm: results of a population screening program. J Vasc Surg. 2003 Jul;38(1):72-7. doi: 10.1016/s0741-5214(03)00135-6. PMID 12844092
- [Background] Vardulaki KA, Walker NM, Couto E, Day NE, Thompson SG, Ashton HA, Scott RA. Late results concerning feasibility and compliance from a randomized trial of ultrasonographic screening for abdominal aortic aneurysm. Br J Surg. 2002 Jul;89(7):861-4. doi: 10.1046/j.1365-2168.2002.02133.x. PMID 12081734
- [Background] Ashton HA, Buxton MJ, Day NE, Kim LG, Marteau TM, Scott RA, Thompson SG, Walker NM; Multicentre Aneurysm Screening Study Group. The Multicentre Aneurysm Screening Study (MASS) into the effect of abdominal aortic aneurysm screening on mortality in men: a randomised controlled trial. Lancet. 2002 Nov 16;360(9345):1531-9. doi: 10.1016/s0140-6736(02)11522-4. PMID 12443589
- [Background] Lindholt JS, Juul S, Henneberg EW. High-risk and low-risk screening for abdominal aortic aneurysm both reduce aneurysm-related mortality. A stratified analysis from a single-centre randomised screening trial. Eur J Vasc Endovasc Surg. 2007 Jul;34(1):53-8. doi: 10.1016/j.ejvs.2006.12.031. Epub 2007 Feb 28. PMID 17331750
- [Background] Davis M, Harris M, Earnshaw JJ. Implementation of the National Health Service Abdominal Aortic Aneurysm Screening Program in England. J Vasc Surg. 2013 May;57(5):1440-5. doi: 10.1016/j.jvs.2012.10.114. Epub 2013 Mar 21. PMID 23523277
- [Background] Baron-Epel O, Keinan-Boker L, Weinstein R, Shohat T. Persistent high rates of smoking among Israeli Arab males with concomitant decrease among Jews. Isr Med Assoc J. 2010 Dec;12(12):732-7. PMID 21348400